

## Università degli Studi di L'Aquila



#### MODULO DI CONSENSO INFORMATO

TITOLO DELLO STUDIO: Studio clinico "No-Profit" per il miglioramento della pratica clinica, per valutare l'efficacia di anakinra nella riduzione dell'emoglobina glicata in soggetti con artrite reumatoide e diabete. Studio randomizzato, controllato, in aperto, per gruppi paralleli.

CODICE DELLO STUDIO: Anakin-RA-Diabetes

| DATA E VERSIONE DELLO STUDIO: Versione Finale del 15/11/12 |
|------------------------------------------------------------|
| CENTRO N.: |
| J. DI ARRUOLAMENTO: |
| NIZIALI DEL PAZIENTE: |
| DELIBERA APPROVAZIONE PARERE C.E. N |
| o sottoscritto (nome e cognome) |
| tà; sesso M F ; data di nascita/_/_ |
| ndirizzo: Via/Piazza |
| CAP Città tel |

#### Dichiaro di:

- partecipare volontariamente allo studio "STUDIO CLINICO "NO-PROFIT" PER IL MIGLIORAMENTO DELLA PRATICA CLINICA, PER VALUTARE L'EFFICACIA DI ANAKINRA NELLA RIDUZIONE DELL'EMOGLOBINA GLICATA IN SOGGETTI CON ARTRITE REUMATOIDE E DIABETE; STUDIO CLINICO RANDOMIZZATO, CONTROLLATO, IN APERTO, PER GRUPPI PARALLELI", avente lo scopo di verificare se la somministrazione di anakinra in pazienti affetti da artrite reumatoide, e da diabete di tipo 2 come comorbidità, è in grado di determinare un miglioramento del controllo glicemico, oltre che dei segni e sintomi dell'AR.
- aver ricevuto dal Medico su menzionato tutte le informazioni chiare ed esaurienti sulle finalità e le procedure dello studio clinico a cui mi è stato chiesto (al mio tutelato) di prendere parte;
- aver letto e compreso il foglio di informazioni che mi è stato consegnato con sufficiente anticipo e che conferma quanto mi è stato verbalmente detto;
- aver avuto l'opportunità di porre domande chiarificatrici e di aver avuto risposte soddisfacenti, come pure di aver avuto la possibilità di informarmi sui particolari dello studio con persona di mia fiducia;
- essere stato/a informato/a sui risultati che potrei trarre (mio tutelato) e sui rischi o disagi ragionevolmente prevedibili, e di aver avuto il tempo sufficiente per decidere;

| Anakin-RA-Diabetes |
|-------------------------------------|
| <i>Versione Finale del 15/11/12</i> |
| Firma Paziente |



## Università degli Studi di L'Aquila



| • | accons | entir | re/non ac | consentire a ch | e lo | sperime | entatore o | il me | dico sopra | menzio | onato invii | una |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | nota, | il | foglio | informativo | al | mio | medico | di | fiducia | nella | persona | di |
| | | | | | | _ circa | la partecip | azion | e a questo | studio c | elinico; | |

- essere consapevole:
  - che la partecipazione allo studio è volontaria e che posso ritirarmi (mio tutelato) dallo studio di mia (sua) spontanea volontà senza fornire giustificazioni, avendo ricevuto la certezza che sia il rifiuto a partecipare allo studio sia il mio eventuale ritiro non influiranno nel ricevere la terapia più idonea al mio (suo) caso;
  - che i miei dati clinici potranno essere esaminati o utilizzati per pubblicazioni scientifiche ma resteranno strettamente riservati nel rispetto della normativa vigente e successive modifiche ed integrazioni;
  - che il Comitato Etico di questa Azienda USL (di cui ho ricevuto il recapito) ha approvato il protocollo sperimentale dello studio;
  - che sarò messo al corrente, del corso della sperimentazione, di qualsiasi nuovo dato possa compromettere la sicurezza del farmaco e la metodica dei trattamenti;
  - del mio diritto ad avere libero accesso alla documentazione relativa alla sperimentazione (assicurativa, clinico-scientifica, farmaco-terapeutica) ed alla valutazione espressa dal Comitato Etico, cui potrò rivolgermi se lo riterrò opportuno;
- che è stata stipulata una Polizza Assicurativa in favore dei soggetti che partecipano allo studio per eventuali danni con la Società Assicuratrice HDI-Garling per indennizzo massimale pari a: € 1.000.000,00 per paziente;
- di dover firmare (io e/o il mio tutelato) due moduli identici del presente consenso informato: un originale verrà trattenuto dal medico (e conservato per almeno 15 anni) e il secondo mi verrà consegnato;
- che per ogni problema o per eventuali informazioni dovrò rivolgermi a:
   Prof. Roberto Giacomelli,
   U.O.C di Reumatologia, Ospedale Civile San Salvatore, via Vetoio, 67100 L'Aquila
   Tel: 0862433395
- che nel mio proprio interesse lo sperimentatore potrà decidere il mio ritiro dallo studio. Pertanto acconsento liberamente alla partecipazione (del mio tutelato) allo studio clinico. La firma su questo modulo non verrà ad incidere sui miei diritti legali (del mio tutelato).

| Letto e approvato (scritto a mano) |
|----------------------------------------------------------------|
| (luogo e data) |
| FIRMA DEL/DELLA PAZIENTE |
| COGNOME E NOME DELL'EVENTUALE RAPPRESENTANTE LEGALMENTE |
| RICONOSCIUTO |
| Anakin-RA-Diabetes Versione Finale del 15/11/12 Firma Paziente |



# Università degli Studi di L'Aquila



### MODULO DI CONSENSO INFORMATO SCRITTO

TITOLO DELLO STUDIO: Studio clinico "No-Profit" per il miglioramento della pratica clinica, per valutare l'efficacia di anakinra nella riduzione dell'emoglobina glicata in soggetti con artrite reumatoide e diabete. Studio clinico randomizzato, controllato, in aperto, per gruppi paralleli.

| CODICE DELLO STUDIO: Anakin-RA | A-Diabetes |
|---|---|
| DATA E VERSIONE DELLO STUDIO | 9: Versione Finale del 15/11/12 |
| CENTRO N: | |
| N.°DI ARRUOLAMENTO: | |
| INIZIALI DEL PAZIENTE: | |
| PAGINA N. DI NN. PAGINE: | |
| COGNOME E NOME DEL MEDICO S | SPERIMENTATORE: |
| OSPEDALE: | |
| FIRMA DELL'EVENTUALE RAPPRE | ESENTANTE LEGALMENTE RICONOSCIUTO |
| Per il testimone imparziale: | |
| Io sottoscritto | dichiaro che il Dott./Prof. |
| ha diffusamente spiegato al Sig./Sig.ra _ | (tutore di) |
| le caratteristiche dello studio sperime | entale in oggetto, secondo quanto riportato nella sche |
| informativa qui allegata, e che lo/a stess | so/a, ha avuto la possibilità di fare tutte le domande che |
| | urientemente informato e quindi ha liberamente accettato |
| aderire allo studio. | |
| FIRMA DEL TESTIMONE IMPARZIA | ALE |

Anakin-RA-Diabetes Versione Finale del 15/11/12 Firma Paziente